CLINICAL TRIAL: NCT02512211
Title: Spanish Validation of "Haemophilia Activities List" (HAL) and "Specific Sport Scale" (HEP-Test-Q) Questionnaires
Brief Title: Validation of Questionnaires HAL and HEP
Acronym: VALIDATION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, PhD, Universidad Católica San Antonio de Murcia
Other Study IDs: VALIDATION; VALIDATION
Record Dates: First submitted 2014-07-22; First posted 2015-07-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Haemophilia
Keywords: Hemophilia; Validation; Questionnaires; Activities; Sport; Patients
MeSH Terms: conditions — Hemophilia A; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients adults: Sample of patients with haemophilia over 18 years of age that will participate in piloting of reliability and validity of the Spanish version of the HAL and HEP questionnaires
- Children with haemophilia: Sign hemophilia patients under 18 years of age that will participate in piloting of reliability and validity of the Spanish version of the HAL and HEP questionnaires
- Parents of children with haemophilia: Sample of parents of children with hemophilia under 18 years of age that will participate in piloting of reliability and validity of the Spanish version of the HAL and HEP questionnaires

SUMMARY:
Spanish Validation of HAL and HEP questionnaire by double translation (English-Spanish-English), with a pilotage pediatric patients with hemophilia and adults and parents of children with hemophilia. The final validity will be obtained with a sample of 60-100 patients with hemophilia

DETAILED DESCRIPTION:
Validation of the Spanish hemophilia specific questionnaires: HAL and HEP (adult version version version children and parents). To do this, there will be a double inverse translation, a pilotage of validity and clarity with a small sample of subjects and analysis of reliability and validity with more than 100 patients and parents of children with hemophilia to complete the validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A and B
* Parents of children with hemophilia A and B, under 18
* Patients who have previously signed the informed consent document

Exclusion Criteria:

* Patients with other congenital coaghulopatías (eg, Von Willebrand's disease)
* Patients with cognitive impairment, or oral or written understanding

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia and parents of children with hemophilia around the country that will participate in study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Translation of the original questionnaire (English) to Spanish | 1 day (Screening visit)
  Three health experienced in the treatment of hemophilia and knowledge of English, translated into Spanish the HAL and HEP questionnaire.
  Two native speakers (English and Spanish), reverse-translate the original text of the HAL and HEP questionnaires and the text translated by the Spanish health
the translated version of the questionnaire | 1 day (Screening visit)
  5 patients with hemophilia under 16, 5 patients with hemophilia adults , and 5 parents of children with hemophilia enrolled randomly will participate in the pilotage.
  The clarity of the questions in Spanish translated version and the relevance of each of the items of the questionnaires will be evaluated.
Sending the questionnaire to a large sample of patients for final validation | 1 day (Screening visit)
  40 hemophilia patients under 16 years old, 60 adult patients with hemophilia and 60 parents of children with hemophilia will participate in the pilotage.
  The validity and reliability of the Spanish version translated from the questionnaires will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: RUBEN CUESTA-BARRIUSO, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (2):
- Spain (2):
  - Universidad de Murcia, Murcia, Murcia
  - Universidad Católica San Antonio, Murcia, Murcia, Murcia